CLINICAL TRIAL: NCT00349245
Title: A Randomized, Double-Blind Comparison Of Dexmedetomidine And Remifentanil For Sedation During Awake Fiberoptic Intubations
Brief Title: Dexmedetomidine vs. Remifentanil for Sedation During AFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Carin A. Hagberg, Professor and Chairman, Joseph C. Gable, MD Endowed Chair, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HSC-MS-06-0173
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Intubation, Endotracheal
Keywords: Endotracheal; Awake fiberoptic intubation; Dexmedetomidine; Remifentanil
MeSH Terms: interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Remifentanil
Drug: Dexmedetomidine

SUMMARY:
The objective of this study is to determine the efficacy and safety of Dexmedetomidine, a selective alpha-2 adrenoceptor agonist, which has recently gained increased popularity for ICU and intraoperative sedation as a sedative during awake fiberoptic intubation, as compared to Remifentanil.

The hypothesis is that Dexmedetomidine will provide at least equal if not better conditions (sedation and analgesia) required for awake fiberoptic intubation (Ramsay Sedation Scale 3) with less respiratory and cardiovascular adverse effects, as well as less recall than Remifentanil.

DETAILED DESCRIPTION:
Awake nasal or oral fiberoptic intubation remains the method of choice for airway management in the expected difficult airway. This technique requires that a patient be comfortable, relaxed, cooperative and able to maintain their airway with spontaneous ventilation.

In order to achieve these conditions, the pharmacologic agent chosen for sedation should be short acting and highly titratable, provide the required amount of sedation and have little suppression of spontaneous ventilation. There have been numerous reports of the use of Remifentanil and Propofol used either alone or in combination to achieve this level of sedation.

Remifentanil has the following advantages which makes it a useful drug for this purpose:

1. Ultra short acting with a constant half life
2. Anti-tussive effects which help prevent coughing with tracheal manipulation
3. Reversible with an antagonist naloxone
4. Attenuates cardiovascular responses to laryngoscopy

Shortcomings of Remifentanil include undesirable side effects, such as hemodynamic instability and respiratory depression.

Dexmedetomidine is a centrally acting, selective alpha-2 agonist which has gained increasing popularity since 1999 as a drug for sedation in ICU settings. It has also been used for intraoperative sedation during surgery under regional anesthesia and for awake craniotomies, as well as for sedation of pediatric patients in different settings. Finally, there are also case reports of Dexmedetomidine being used for awake fiberoptic tracheal intubation.

Theoretically, the pharmacokinetic and pharmacodynamic properties of Dexmedetomidine make it an ideal drug as a single agent for sedation for awake fiberoptic intubation. Venn et al showed that in both healthy individuals and ICU patients, Dexmedetomidine shows a rapid onset and equally rapid distribution half life with quick recovery. This study also demonstrated stable hemodynamics during airway manipulation (extubation) with no adverse cardiovascular or respiratory events during the study.

Other studies have demonstrated that Dexmedetomidine attenuates cardiovascular responses to laryngoscopy and intubation and reduces the need for perioperative opioids. In small doses, it has been demonstrated to have good sedative, amnestic and analgesic effects, as well as anti-sialogogue effects.

Dexmedetomidine does, however, have some drawbacks. In higher bolus doses it can cause hemodynamic changes, such as excessive bradycardia and hypertension followed by hypotension. This drug has also been associated with decreased regional and global cerebral blood flow despite maintenance of MAP within the auto-regulating parameters. These deleterious effects are more prominent in patients with hypovolemia, systemic vasoconstriction, AV block and with rapid bolus infusion.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent must be obtained after the nature of the study has been fully explained.
* Patients undergoing any procedure requiring general anesthesia with an endotracheal tube.
* Patients that have been assessed by an attending anesthesiologist to have an airway requiring awake fiberoptic intubation.
* Adult patients > 18 yrs. old, ASA I - III.

Exclusion Criteria:

* Patients expected to have severe adverse side effects to Dexmedetomidine including:

  1. Previous allergy to the drug.
  2. 3rd degree AV Block
  3. Hypovolemic hypotension
  4. Systemic vasoconstriction
* Patients expected to have a severe adverse side effect to Remifentanil. This includes:

  1. Previous allergy to the drug.
  2. Patients suspected of being overly sensitive to narcotics.
* Patients with significant cardiovascular disease or ASA physical status IV and V

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Patient's reaction to procedure, as it occurs, ie. grimace, gag, verbalized pain. | duration of intubation
Memory recall | post operative, immediately every 30 min for 3 hours and 24 hours

SECONDARY OUTCOMES:
NIBP | duration of intubation and first 15 minutes of surgery
HR | duration of intubation and first 15 minutes of surgery
Cardiac rhythm | duration of surgery
Oxygen saturation | duration of intubation and first 15 minutes of surgery
End-tidal carbon dioxide | duration of intubation and first 15 minutes of surgery
Continuous ECG | duration of intubation and first 15 minutes of surgery
Pulse oximetry | duration of intubation and first 15 minutes of surgery
Bispectral index | duration of intubation
Respiratory rate | duration of intubation and first 15 minutes of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carin A Hagberg, M.D., Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States